CLINICAL TRIAL: NCT00005288
Title: Epidemiology and Pulmonary Response To Organic Dust Exposure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2009
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2001-04

CONDITIONS: Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To characterize the nature of pulmonary responses to organic dust exposures in order to gain insight into patterns of respiratory disease in agricultural workers.

DETAILED DESCRIPTION:
BACKGROUND:

In 1986 when the study began, agriculture was one of the largest employers in the United States, comprising nearly 12 million people. Farm workers were hospitalized more frequently than other occupational groups and were found to have the highest number of restricted activity days due to injury and illness. Much of this was due to frequent and disabling farm related accidents which made agriculture the most hazardous occupation in the United States. Agricultural workers were also found to have high rates of respiratory disability, compared with other industrial sectors, based on Social Security disability records.

The common denominator for respiratory disorders among agricultural workers was exposure to organic dust which was recognized to be a complex mixture of vegetable particles and fragments, microorganisms and their products, insects and insect fragments, feed additives including fish meal and antibiotics, and avian and rodent proteins. While the vegetable dust itself was by far the most important exposure, individual circumstances of growing, storage and subsequent use of the product from which the organic dust arose, influenced specific exposures. In certain situations, like animal confinement housing, irritant gases including ammonia and hydrogen sulfide co-existed with an organic dust to further vary respiratory exposure.

Workers exposed in Iowa swine production units were known to be significantly exposed to grain dust, endotoxin, animal danders and other proteins, ammonia and hydrogen sulfide gas, and a variety of microorganisms including fungi and thermophilic actinomycetes. Cross-sectional epidemiological surveys had documented a high prevalence of respiratory symptoms including chronic cough, phlegm and wheezing, but also prominent constitutional symptoms including fever, myalgias and malaise. This study was one of several projects supported by a Specialized Center of Research in Occupational and Immunologic Lung Disease.

Funding represents approximately 35 percent of the dollars of the Specialized Center of Research in Occupational and Immunologic Lung Disease (P50HL37121) used to support epidemiologic studies.

DESIGN NARRATIVE:

A nested case-control study was carried out on a previously studied cohort. Members of the cohort were resurveyed in the first year of the study. All participants received a routine physical examination, chest x-ray, electrocardiogram if over 40 years of age, routine laboratory tests, methacholine challenge, intradermal skin testing, and bronchoalveolar lavage. Cases for the swine confinement farmer cohort were selected if they had FEF50 of 60 percent or less of predicted for age, sex, height, and race. Three referents for each case were randomly selected from all swine confinement farmers not selected as cases, non-confinement farmers, and blue collar workers. Measurements were repeated in the fourth year, finishing in the fifth year of the study. The study determined: the extent to which epidemiological studies underestimated pulmonary responses and impairments among agricultural workers; the environmental risk factors significantly related to cases; whether atopy and heightened airway reactivity were significantly associated risk factors. The subproject was not renewed in 1992.

The study completion date listed in this record was obtained from the "End Date" entered in the old format Protocol Registration and Results System (PRS).

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-12; Study Completion 1991-11 (Actual)

REFERENCES:
- [Background] Merchant JA: Agricultural Respiratory Disease, In: Seminars in Respiratory Medicine - Vol. 7, Number 3. Thieme Inc, pp 211-224, New York, 1986
- [Background] Merchant JA: Silicosis Issues - Past, Present, Future. Published in Book: Silica, Silicosis, and Cancer: Controversy in Occupational Medicine, 1986, Goldsmith DF, Winn DM, Shy CM (Eds), Praeger Special Studies, Praeger Scientific, pp 87-90, New York, 1986
- [Background] Omenn GS, Merchant J, Boatman E, Dement JM, Kuschner M, Nicholson W, Peto J, Rosenstock L. Contribution of environmental fibers to respiratory cancer. Environ Health Perspect. 1986 Dec;70:51-6. doi: 10.1289/ehp.867051. PMID 3830113
- [Background] Merchant JA. Preparing for disaster. Am J Public Health. 1986 Mar;76(3):233-5. doi: 10.2105/ajph.76.3.233. No abstract available. PMID 3946707
- [Background] Merchant JA: Contribution to Report The Health Consequences of Smoking: Cancer and Chronic Lung Disease in the Workplace: A Report of the Surgeon General. U.S. Department of Health and Human Services, Public Health Service, Office on Smoking and Health, U.S. Government Printing Service, Washington, D.C., 1986
- [Background] Merchant JA, Boehlecke BA, Taylor G (EDs): Occupational Respiratory Diseases, U.S. Department of Health and Human Services, Public Health Service, Centers for Disease Control, National Institute for Occupational Safety and Health, U.S. Government Printing Office, Washington, D.C., 1986
- [Background] Dement JM, Merchant JA: Chapter III. C: Asbestosis, in Occupational Respiratory Diseases, U.S. Department of Health and Human Services, Public Health Service, Centers for Disease Control, National Institute for Occupational Safety and Health, U.S. Government Printing Office, Washington, D.C., 1986
- [Background] Merchant JA: Chapter VI. Byssinosis, in Occupational Respiratory Diseases, U.S. Department of Health and Human Services, Public Health Services, Centers for Disease Control, National Institute for Occupational Safety and Health, U.S. Government Printing Office, Washington, D.C., 1986
- [Background] Merchant JA, Hodous T, Taylor G, Reger R: Chapter III. D: Coal Workers Pneumoconiosis, in Occupational Respiratory Diseases, U.S. Department of Health and Human Services, Public Health Service, Centers for Disease Control, National Institute for Occupational Safety and Health, U.S. Government Printing Office, Washington, D.C., 1986
- [Background] Merchant JA. New dimensions in occupational medicine. Iowa Med. 1987 Apr;77(4):177-9. No abstract available. PMID 3583660
- [Background] Merchant JA. Agricultural exposures to organic dusts. Occup Med. 1987 Apr-Jun;2(2):409-25. PMID 3303387
- [Background] Muldoon JT, Wintermeyer LA, Eure JA, Fuortes L, Merchant JA, Van Lier SF, Richards TB. Occupational disease surveillance data sources, 1985. Am J Public Health. 1987 Aug;77(8):1006-8. doi: 10.2105/ajph.77.8.1006. PMID 3605466
- [Background] Merchant JA, Donham KJ: Health Risks from Animal Confinement Units. Proceedings of the International Symposium on Health and Safety in Agriculture. Saskatoon, Canada. In press, 1987
- [Background] Guernsey JR, Morgan DP, Marx JJ, Horvath EP, Pierce P, Merchant JA: The Prognostic Significance of Farmer's Lung Disease Antibodies Relative to Measures of Respiratory Disease. Proceedings of the International Symposium on Health and Safety in Agriculture, Saskatoon, Canada. In press, 1987
- [Background] Leistikow BN, Donham KJ, Merchant JA: Health Hazards of Poultry Production: Proceedings of the International Symposium on Health and Safety in Agriculture, Saskatoon, Canada. In press, 1987
- [Background] Twiggs JT, Gray RL, Marx JJ Jr. House dust mite (Dermatophagoides farinae) allergen levels in three different sources from homes of patients with allergy to house dust mite. Clin Rev Allergy. 1988 Spring;6(1):35-43. doi: 10.1007/BF02914980. No abstract available. PMID 3383075
- [Background] Merchant JA: Occupational Parenchymal Lung Disease. Kelley: Textbook of Internal Medicine. In press, 1988
- [Background] LaMarte FP, Merchant JA, Casale TB. Acute systemic reactions to carbonless copy paper associated with histamine release. JAMA. 1988 Jul 8;260(2):242-3. PMID 2455072
- [Background] Schwartz DA, Galvin JR, Dayton CS, Stanford W, Merchant JA, Hunninghake GW. Determinants of restrictive lung function in asbestos-induced pleural fibrosis. J Appl Physiol (1985). 1990 May;68(5):1932-7. doi: 10.1152/jappl.1990.68.5.1932. PMID 2361895
- [Background] Donham KJ, Merchant JA, Lassise D, Popendorf WJ, Burmeister LF. Preventing respiratory disease in swine confinement workers: intervention through applied epidemiology, education, and consultation. Am J Ind Med. 1990;18(3):241-61. doi: 10.1002/ajim.4700180303. PMID 2220828
- [Background] Merchant JA, Donham KJ, Popendorf WJ, Burmeister LF, Lassise DG, Lee NF, Weinrich AJ: Acute Responses Among Swine Confinement Workers. Proceedings of Agricultural, Occupational, and Environmental Health: Health Policy Strategies for the Future. Iowa City, Iowa. In press 1988
- [Background] Schwartz DA, Landas SK, Lassise DL, Burmeister LF, Hunninghake GW, Merchant JA. Airway injury in swine confinement workers. Ann Intern Med. 1992 Apr 15;116(8):630-5. doi: 10.7326/0003-4819-116-8-630. PMID 1546862
- [Background] Marx JJ Jr, Twiggs JT, Ault BJ, Merchant JA, Fernandez-Caldas E. Inhaled aeroallergen and storage mite reactivity in a Wisconsin farmer nested case-control study. Am Rev Respir Dis. 1993 Feb;147(2):354-8. doi: 10.1164/ajrccm/147.2.354. PMID 8430958